CLINICAL TRIAL: NCT03277950
Title: Effect of Game-based Virtual Reality Training on Upper Extremity Movement in Individuals With Subacute Stroke
Brief Title: Effect of Virtual Reality Game on Upper Limb Movement in Individuals With Stroke
Acronym: VRULS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vimonwan Hiengkaew (Other)
Responsible Party: Sponsor-Investigator, Vimonwan Hiengkaew, Associate professor, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/097.0906
Record Dates: First submitted 2017-08-27; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Stroke; Movement, Abnormal
Keywords: virtual reality; feedback
MeSH Terms: conditions — Stroke; Dyskinesias

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality with feedback (Experimental): Participants received training via virtual reality game with feedback, 60 minutes/day, 3 days/week for 4 weeks, then follow up after 4 weeks.
  Interventions: Other: Virtual reality with feedback
- virtual reality without feedback (Active Comparator): Participants received training via virtual reality game without feedback, 60 minutes/day, 3 days/week for 4 weeks, then follow up after 4 weeks.
  Interventions: Other: Virtual reality without feedback
- Healthy (Other): Participants do not play virtual reality game.
  Interventions: Other: Healthy

INTERVENTIONS:
Other: Virtual reality with feedback — Individuals with stroke play game with correction of movement.
  Arms: virtual reality with feedback
Other: Virtual reality without feedback — Individuals with stroke play game without correction of movement.
  Arms: virtual reality without feedback
Other: Healthy — Healthy do not play game
  Arms: Healthy

SUMMARY:
Individuals with stroke show abnormal movement pattern of upper limb. The movement pattern needs to be corrected. There are several methods to train normal movement. Exercise with technology is an active movement and affects sensory and cognitive systems. It may benefit to individuals with stroke in training.

DETAILED DESCRIPTION:
Individuals with stroke sign informed consent. They are trained with virtual reality game with and without feedback from a researcher. Age-matched healthy play the same game as individuals with stroke do. Both individuals with stroke and healthy are measured upper limb movement pattern.

ELIGIBILITY:
Inclusion Criteria:

Individuals with stroke

1. 45 - 65 years old
2. First ischemic or hemorrhagic stroke
3. Right hemiparesis
4. Right dominant handedness
5. Within 6 months after stroke
6. Discharge from hospital and stay at home
7. Normal dynamic sitting balance
8. At least 120 degrees of shoulder flexion and 45 degrees of shoulder extension by passive range of motion
9. Active movement at least stage 3 by Chedoke-McMaster Stroke Assessment
10. Muscle tone graded 1-2 by Modified Ashworth Scale in 2 of 3 muscle groups including shoulder adductor, internal rotator or/and elbow flexor groups
11. No cognitive impairment

Healthy individuals

1. Have same gender and age within range of ±5 years of individuals with stroke
2. Right handedness
3. Active range of motion of shoulder flexion and extension at least 120°and 45° respectively
4. No cognitive impairment

Exclusion Criteria:

Individual with stroke and healthy

1. Have cyber-sickness
2. Obesity
3. Ataxic movement
4. Loss visual field or visual neglect
5. Loss exteroceptive sensation
6. Impaired or loss proprioceptive sensation
7. Receive the occupation therapy on upper extremity
8. Muscle contracture at the scapula, shoulder and elbow
9. Pain at the scapula, shoulder and elbow
10. History of fracture or surgery at head, shoulder, scapula, and elbow
11. Shoulder subluxation
12. Other neurological disorders
13. Uncontrolled hypertension
14. Myocardial infarction
15. Seizure or epilepsy
16. Pacemaker or hemodialysis vascular access

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2018-09-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
kinematic data | 10 minutes
  angle of shoulder, elbow, and forearm

SECONDARY OUTCOMES:
Upper limb performance | 10 minutes
  doing task according to Fugl Mayer
muscle tone | 2 minutes
  assessing muscles of shoulder, elbow, and forearm according to Modified Ashworth Scale

CONTACTS AND LOCATIONS:
Overall Officials: Vimonwan Hiengkaew, PhD, Study Chair — Mahidol University; Peemonkong Wattananon, PhD, Study Director — Mahidol University; Sirada Lolak, BSc, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No